CLINICAL TRIAL: NCT03549130
Title: Pivotal Subjective Sleep Study of a Nasal Dilator
Brief Title: A Pivotal Study to Assess the Effectiveness of Nasal Dilator (Breathe Right Nasal Strips)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202246; B3570877 (Other: GSK other Identifier)
Record Dates: First submitted 2018-05-25; First posted 2018-06-07 (Actual); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Congestion, Nasal
MeSH Terms: conditions — Nasal Obstruction | interventions — Culture Media

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active nasal strip group (Experimental): Participants of this treatment arm applied sufficient quantity of commercially available nasal strips (small/medium size) outside of the nose, from alar crease to alar crease, as per dispensing instructions
  Interventions: Device: Breathe Right Tan (small/medium) nasal strips
- Placebo nasal strip group (Placebo Comparator): Participants of this treatment arm applied sufficient quantity of Asymmetric Butterfly Placebo ABP-NH Nasal Strips (small/medium size) outside of the nose, from alar crease to alar crease, as per dispensing instructions
  Interventions: Other: Placebo nasal strip

INTERVENTIONS:
Device: Breathe Right Tan (small/medium) nasal strips — Participants of this treatment arm applied sufficient quantity of commercially available nasal strips (Breathe Right Tan), small/medium sized outside of the nose, from alar crease to alar crease, as per dispensing instructions, prior to sleeping. Participants used their assigned strip every night, for approximately 8 hours, but no more than 12 hours per night, for two weeks
  Arms: Active nasal strip group
Other: Placebo nasal strip — Participants of this treatment arm applied sufficient quantity of Asymmetric Butterfly Placebo ABP-NH Nasal Strips, small/medium sized outside of the nose, from alar crease to alar crease, as per dispensing instructions, prior to sleeping. Participants used their assigned strip every night, for approximately 8 hours, but no more than 12 hours per night, for two weeks
  Arms: Placebo nasal strip group

SUMMARY:
This randomized, double-blind, parallel group, placebo-controlled study assessed subjective measures of nasal airway breathing immediately after application in the morning upon awakening after use of breathe right nasal strips (BRNS). Participants who met the entrance criteria, were currently suffering from nasal congestion, reported trouble with their sleep and had baseline nasal openness scores at bedtime during the qualification phase of ≤ 70 on a 100-point Visual Analogue Scale (VAS) on at least four of seven qualification nights were randomized to one of two treatments for use at home. Participants returned to the study site after 7 and 14 days of nightly nasal strip use, respectively. At the two return visits, a validated subjective questionnaire, the Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ), measured response.

DETAILED DESCRIPTION:
The study had a screening phase, a one-week baseline qualification and a two-week treatment phase. Participants who met the entrance criteria, who were currently suffering from nasal congestion every night or almost every night, reported trouble with their sleep and had baseline nasal openness scores at bedtime during the qualification phase of ≤ 70 on a 100-point VAS on at least four of seven qualification nights were randomized to one of two treatments for use at home. During the two-week in-home treatment phase, daily diaries measuring the perception of nasal breathing and nasal congestion using a VAS were completed. Participants returned to the study site after 7 and 14 days of nightly nasal strip use, respectively. At the two return visits, a validated subjective questionnaire, the NRQLQ, measured response.

ELIGIBILITY:
Inclusion Criteria:

* Consent: Demonstrated understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Compliance: Understands and is willing, able and likely to comply with all study procedures and restrictions.
* General Health: Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination.
* Contraception: Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception.
* Leptorrhine Nose: Has a leptorrhine nose as defined in Appendix I to this protocol (nasal tip protrusion index of 45 or greater)
* Chronic Nasal Congestion: Complains of chronic nocturnal nasal congestion for at least the last year. When experiencing nasal congestion, complains always or almost always every night.
* Sleep: Reports trouble with sleep.
* VAS Nasal Openness Qualifying Question: Has baseline nasal openness scores at bedtime during the one-week baseline qualification phase of ≤ 70 on a 100-point VAS where 0=extremely blocked and 100=extremely open on at least four of seven nights.

Exclusion Criteria:

* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds), allergy or atopic reaction to adhesive bandages or latex.
* Participant has current or a history of skin cancer, chronic skin condition, or eczema on the face or nose.
* Participant has visible open sores, sunburn, irritation on the face or nose immediately prior to randomization.
* Participant has been diagnosed with sleep apnea in a sleep laboratory.
* Participant has had a diagnosis of another major sleep disorder (i.e. primary insomnia, i.e. regularly sleeping less than six hours per night, sleep insufficiency, i.e. sleeping >two hours more on non-work days as compared to work days, narcolepsy, restless leg syndrome, or periodic limb movement disorder).
* Participant has a non-typical sleep schedule (e.g. shift-work).
* Participant plans travel involving time-zone changes during the study period.
* Regular/habitual consumption of more than five cups or glasses per day of xanthine-containing beverages (i.e. tea, coffee, cola).
* Participant currently uses any product or medication that has an effect on nasal congestion or sleep. Participant must have discontinued use of the following products according to the timings specified below:

  a) Prior to initiation of the baseline qualification phase: i. Use of any substance with psychotropic effects or properties known to affect sleep/wake, including but not limited to: neuroleptics, morphine/opioid derivatives, sedative antihistamines, stimulants, antidepressants, clonidine, barbiturates, anxiolytics, thalidomide, hypnotics and sedatives. Use of over-the-counter (OTC) sleep promoting agents including diphenhydramine, doxylamine, tryptophan, valerian root, kava kava, melatonin, St John's Wort and Alluna. Use of OTC alertness aids including caffeine and guarana.

ii. Lubricating sprays/rinses/throat strips iii. Devices prescribed or used for sleep disordered breathing including Continuous Positive Airway Pressure (CPAP), mandibular advancement devices, tongue displacement devices iv. Use of any intranasally administered medications (e.g. Miacalcin) b) Within 3 days prior to the initiation of the baseline qualification phase: i. Oral decongestants ii. Short-acting prescription and non-prescription antihistamines, including ocular preparations and antihistamines contained in OTC sleep medications or 'night time' pain formulations (e.g. Benadryl, Chlortrimeton, Dimetane, Tavist) iii. Intranasal, oral or inhaled anticholinergics (e.g. Atrovent) iv. Long-acting beta agonists (e.g. Serevent) v. Oral antileukotrienes c) Within 7 days prior to the initiation of the baseline qualification phase: i. Any topical nasal decongestants (nasal sprays, drops, etc). ii. OTC products such as chin straps, pillows, internal/external nasal dilators.

d) Within 10 days prior to initiation of the baseline qualification phase: i. Long-acting antihistamines (e.g. Allegra, Claritin, Clarinex, Zyrtec). e) Within 14 days prior to initiation of the baseline qualification phase: i. Intranasal cromolyn ii. Intranasal antihistamines (e.g. Astelin, Astepro) f) Within 4 weeks prior to the initiation of the baseline qualification phase: i. Intranasal corticosteroids g) Within 8 weeks prior to the initiation of the baseline qualification phase: i. Inhaled oral, intramuscular, intravenous, ocular and/or dermatological corticosteroid (with the exception of 1% or less topical hydrocortisone products) h) Within 3 months prior to the baseline qualification phase: i. Intranasal vaccines.

* Participant has experienced an acute upper respiratory tract infection during the qualification phase and/or at the Baseline visit.
* Participant abuses alcohol (regularly drinks more than 3 drinks per day) or has a recent history (within last 2 years) of substance or alcohol abuse
* Participant has a positive urine drug screening result (dipstick) for drugs of abuse (cannabinoids, opiates, amphetamines, methamphetamine, cocaine, barbiturates, methadone and/or its metabolites, ecstasy).
* Participant has self-reported severe, unstable disease states (e.g. myocardial infarction, congestive heart failure, diabetes, cirrhosis, cancer, epilepsy, or stroke), pain syndromes, (e.g. fibromyalgia) or any medical or surgical condition that places the Participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study or who in the judgement of the principal investigator would not be suitable for entry into this study.
* Severe nasal obstruction caused by structural abnormality that renders the Participant unsuitable for the study in the opinion of the investigator, i.e. significant nasal polyps, severe deviated septum.
* Participant who is pregnant or nursing, by self-report.
* Participation in another clinical study.
* Receipt of an investigational drug within 30 days of the start of the baseline qualification phase.
* Previous participation in this study.
* Personnel: An employee of the sponsor or the study site or members or their immediate family.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-11-04 (Actual); Primary Completion 2011-02-17 (Actual); Study Completion 2011-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - Concentrics Research, Indianapolis, Indiana
  - TKL Research Inc, Paramus, New Jersey

REFERENCES:
- [Derived] Noss MJ, Ciesla R, Shanga G. Sleep Quality and Congestion with Breathe Right Nasal Strips: Two Randomized Controlled Trials. Adv Ther. 2019 Aug;36(8):1975-1985. doi: 10.1007/s12325-019-01005-5. Epub 2019 Jun 17. PMID 31209698

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at two centers in USA.
Pre-assignment Details: A total of 235 participates were screened, out of which 130 participants were enrolled and randomized in the study. 105 participants were not randomized as 104 of which did not meet study criteria, 1 had adverse event.
Period: Overall Study
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Started | 64 | 66
Completed | 64 | 64
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The ITT (N= 128) population included all participants who were randomized into the study and had at least one post-baseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Customized [Mean (Standard Deviation); unit: Years] | 47.1 (11.27) | 48.4 (13.74) | 47.8 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 92
  Male | 16 | 20 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 55 | 52 | 107
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Average Score of Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) for Each Domain Problems (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) at Day 7
Description: Participants scored all the domains of NRQLQ using same 7 points scales where 0=Not troubled and 6=extremely troubled. Domains: Sleep problems (difficulty getting sleep, unable to get a good night sleep or wake up during the night, restless [tossing and turning] and having to get up because stuffy nose or to blow nose using the score, scores range: Min-Max [0-24]); Sleep time problems (Nasal congestion or stuffy nose, sinus pressure or pain, runny nose, post-nasal drip [drainage down back of nose/throat], and headache, scores range: 0- 30); Symptoms on waking in the morning (Feel tired and unrefreshed, nasal congestion or stuffy nose, congestion in sinuses, takes time to clear nighttime drainage after waking up, scores range:0-24); practical problems (have to avoid symptom triggers (such as dust, cigarette smoke, strong smells and perfumes), need to rub nose or eyes, and have to take medication, scores range: 0-18). Lower scores indicate improvement in the rhinitis symptoms.
Time Frame: At baseline and Day 7
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on Scale
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Number analyzed (Participants) | 64 | 64
Score on Scale
  Sleep Problems | -4.94 [-5.85 to -4.02] | -4.17 [-5.09 to -3.25]
  Sleep Time Problems | -6.30 [-7.46 to -5.14] | -4.51 [-5.67 to -3.34]
  Symptoms on waking in the morning | -6.49 [-7.55 to -5.44] | -4.87 [-5.93 to -3.80]
  Practical problems | -2.98 [-3.70 to -2.27] | -2.28 [-3.00 to -1.56]
Statistical Analysis 1: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for Sleep problems; Test type: Superiority; p = 0.2446, ANCOVA — Between treatment p-values; Treatment,site used as factors;following variables as covariate:baseline, age,level of congestion symptoms at baseline,Berlin score,Epworth sleepiness; Least Square (LS) mean difference = -0.77, 95% CI 2-sided [-2.06 to 0.53] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 2: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for Sleep Time Problems; Test type: Superiority; p = 0.0333, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -1.80, 95% CI 2-sided [-3.45 to -0.14] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 3: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for Symptoms on Waking in the Morning; Test type: Superiority; p = 0.0345, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -1.63, 95% CI 2-sided [-3.13 to -0.12] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 4: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for Practical Problems; Test type: Superiority; p = 0.1711, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.71, 95% CI 2-sided [-1.72 to 0.31] — Difference between treatments of adjusted mean change from baseline

2. Primary Outcome: Change From Baseline in Mean Average Score of Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) for Each Domain Problems (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) at Day 14
Description: as for outcome 1
Time Frame: At Baseline and Day 14
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score On scale
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Number analyzed (Participants) | 64 | 64
Score On scale
  Sleep Problems | -6.34 [-7.31 to -5.36] | -5.87 [-6.85 to -4.89]
  Sleep Time Problems | -7.30 [-8.47 to -6.12] | -6.32 [-7.50 to -5.15]
  Symptoms on Walking in the Morning | -7.25 [-8.28 to -6.23] | -6.54 [-7.56 to -5.52]
  Practical Problems | -3.47 [-4.17 to -2.77] | -2.66 [-3.36 to -1.95]
Statistical Analysis 1: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for Sleep problems; Test type: Superiority; p = 0.5063, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.47, 95% CI 2-sided [-1.85 to 0.92] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 2: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for Sleep time problems; Test type: Superiority; p = 0.2496, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.97, 95% CI 2-sided [-2.64 to 0.69] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 3: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for symptoms on waking in the morning; Test type: Superiority; p = 0.3325, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.71, 95% CI 2-sided [-2.16 to 0.74] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 4: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of NRQLQ between active and placebo strip group for practical problems; Test type: Superiority; p = 0.1088, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.81, 95% CI 2-sided [-1.81 to 0.18] — Difference between treatments of adjusted mean change from baseline

3. Primary Outcome: Change From Baseline in Mean Average Score for All the Four Questions of Domain Symptoms on Waking in the Morning of Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire (NRQLQ) at Day 7
Description: Participants scored for domain Symptoms on waking in the morning of NRQLQ using 7 points scale: 0=not troubled, 1=hardly troubled at all, 2=somewhat troubled, 3= moderately troubled, 4=quite a bit troubled, 5=very troubled, 6=extremely troubled. Questionnaire for this domain included: Feel tired and unrefreshed, nasal congestion or stuffy nose, congestion in sinuses, takes time to clear night time drainage after waking up. Lower scores indicate improvement in the rhinitis symptoms
Time Frame: At Baseline and Day 7
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on Scale
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Number analyzed (Participants) | 64 | 64
Score on Scale
  Feel Tired and Unrefreshed | -1.40 [-1.70 to -1.10] | -1.15 [-1.45 to -0.84]
  Nasal congestion or stuffy nose | -1.71 [-2.00 to -1.43] | -1.34 [-1.63 to -1.05]
  Congestion in sinuses | -1.59 [-1.90 to -1.28] | -1.04 [-1.36 to -0.73]
  Takes time to clear nighttime drainage | -1.80 [-2.13 to -1.47] | -1.33 [-1.66 to -1.00]
Statistical Analysis 1: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of Symptoms on Waking in the Morning in NRQLQ between active and placebo strip group for feel tired and unrefreshed; Test type: Superiority; p = 0.2513, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.25, 95% CI 2-sided [-0.68 to 0.18] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 2: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of Symptoms on Waking in the Morning in NRQLQ between active and placebo strip group for nasal congestion or stuffy nose; Test type: Superiority; p = 0.0743, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.37, 95% CI 2-sided [-0.78 to 0.04] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 3: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of Symptoms on Waking in the Morning in NRQLQ between active and placebo strip group for congestion in sinuses; Test type: Superiority; p = 0.0158, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.55, 95% CI 2-sided [-0.99 to -0.10] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 4: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of Symptoms on Waking in the Morning in NRQLQ between active and placebo strip group for time to clear nighttime drainage after waking up; Test type: Superiority; p = 0.0489, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.47, 95% CI 2-sided [-0.94 to 0.00] — Difference between treatments of adjusted mean change from baseline

4. Primary Outcome: Change From Baseline in Mean Average Score for All the Four Questions of Domain Symptoms on Waking in the Morning of Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire at Day 14
Description: as for outcome 3
Time Frame: At Baseline and Day 14
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on Scale
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Number analyzed (Participants) | 64 | 64
Score on Scale
  Feel Tired and Unrefreshed | -1.65 [-1.92 to -1.39] | -1.46 [-1.72 to -1.20]
  Nasal congestion or stuffy nose | -1.96 [-2.26 to -1.67] | -1.82 [-2.11 to -1.52]
  Congestion in sinuses | -1.71 [-2.00 to -1.42] | -1.70 [-1.99 to -1.41]
  Takes time to clear nighttime | -1.93 [-2.26 to -1.60] | -1.56 [-1.89 to -1.24]
Statistical Analysis 1: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3034, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.19, 95% CI 2-sided [-0.57 to 0.18] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 2: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.4891, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.15, 95% CI 2-sided [-0.57 to 0.27] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 3: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.9498, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.01, 95% CI 2-sided [-0.43 to 0.40] — Difference between treatments of adjusted mean change from baseline
Statistical Analysis 4: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.1235, ANCOVA — Between treatment p-values; [statistical method as in outcome 1, analysis 1]; LS mean difference = -0.36, 95% CI 2-sided [-0.83 to 0.10] — Difference between treatments of adjusted mean change from baseline

5. Primary Outcome: Number of Participants Showing Improvement for Each Domain Problems (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) of Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire at Day 7
Description: Participants scored all the domains of NRQLQ using 7 points scale,0=Not troubled,1=hardly troubled at all,2=somewhat troubled,3=moderately troubled, 4=quite a bit troubled,5=very troubled,6=extremely troubled.Sleep problems (difficulty getting sleep,unable to get good night sleep/wake up during night, restless [tossing and turning],having to get up because stuffy nose or blow nose using score,scores range:Min-Max[0-24]),Sleep time problems(Nasal congestion or stuffy nose,sinus pressure or pain,runny nose,post-nasal drip[drainage down back of nose/throat],headache,scores range:0-30);Symptoms on waking in morning(Feel tired and unrefreshed,nasal congestion/stuffy nose,congestion in sinuses,takes time to clear nighttime drainage after waking up,scores range:0-24);practical problems(have to avoid symptom triggers(such as dust,cigarette smoke,strong smells, perfumes),rub nose/eyes,take medication,score range:0-18).Lower scores relative to baseline indicate improvement in rhinitis symptoms.
Time Frame: At Day 7
Population: The ITT (N= 128) population included all participants who were randomized into the study and had had at least one post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Number analyzed (Participants) | 64 | 64
Participants
  Improvement:all of the items in sleep problems | 20 | 21
  Improvement:any of the items in sleep problems | 59 | 61
  Improvement:all of items in sleep time problems | 21 | 17
  Improvement:any of items in sleep time problems | 58 | 61
  Improvement:all of items in symptom on walking(AM) | 37 | 28
  Improvement:any of items in symptom on walking(AM) | 60 | 58
  Improvement:all of the items in practical problems | 9 | 12
  Improvement:any of the items in practical problems | 53 | 48
Statistical Analysis 1: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in sleep problems; Test type: Superiority; p = 0.8498, Chi-squared — P-value are based on chi-square test
Statistical Analysis 2: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in sleep problems; Test type: Superiority; p = 0.4652, Chi-squared — P-value are based on chi-square test
Statistical Analysis 3: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in sleep time problems; Test type: Superiority; p = 0.4390, Chi-squared — P-value are based on chi-square test
Statistical Analysis 4: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in sleep time problems; Test type: Superiority; p = 0.2997, Chi-squared — P-value are based on chi-square test
Statistical Analysis 5: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in symptoms on waking in AM; Test type: Superiority; p = 0.1116, Chi-squared — P-value are based on chi-square test
Statistical Analysis 6: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in symptoms on waking in AM; Test type: Superiority; p = 0.5101, Chi-squared — P-value are based on chi-square test
Statistical Analysis 7: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in practical problems; Test type: Superiority; p = 0.4740, Chi-squared — P-value are based on chi-square test
Statistical Analysis 8: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in practical problems; Test type: Superiority; p = 0.2787, Chi-squared — P-value are based on chi-square test

6. Primary Outcome: Number of Participants Showing Improvement for Each Domain Problems (Sleep, Sleep Time, Symptoms on Waking in the Morning, and Practical Problems) of Nocturnal Rhinoconjunctivitis Quality of Life Questionnaire at Day 14
Description: as for outcome 5
Time Frame: At Day 14
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
Number analyzed (Participants) | 64 | 64
Participants
  Improvement:all of the items in sleep problems | 31 | 34
  Improvement:any of the items in sleep problems | 59 | 60
  Improvement:all of items in sleep time problems | 24 | 26
  Improvement:any of items in sleep time problems | 60 | 62
  Improvement:all of items in symptom on walking(AM) | 35 | 39
  Improvement:any of items in symptom on walking(AM) | 62 | 63
  Improvement:all of the items in practical problems | 14 | 13
  Improvement:any of the items in practical problems | 55 | 51
Statistical Analysis 1: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in sleep problems; Test type: Superiority; p = 0.5958, Chi-squared — P-value are based on chi-square test
Statistical Analysis 2: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in sleep problems; Test type: Superiority; p = 0.7296, Chi-squared — P-value are based on chi-square test
Statistical Analysis 3: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in sleep time problems; Test type: Superiority; p = 0.7171, Chi-squared — P-value are based on chi-square test
Statistical Analysis 4: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in sleep time problems; Test type: Superiority; p = 0.4030, Chi-squared — P-value are based on chi-square test
Statistical Analysis 5: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in symptoms on waking in AM; Test type: Superiority; p = 0.4741, Chi-squared — P-value are based on chi-square test
Statistical Analysis 6: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in symptoms on waking in AM; Test type: Superiority; p = 0.5591, Chi-squared — P-value are based on chi-square test
Statistical Analysis 7: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on all of the items in practical problems; Test type: Superiority; p = 0.8285, Chi-squared — P-value are based on chi-square test
Statistical Analysis 8: Comparison: Active Nasal Strip Group vs Placebo Nasal Strip Group; Treatment comparison of participants showing improvement based on NRQLQ on any of the items in practical problems; Test type: Superiority; p = 0.3487, Chi-squared — P-value are based on chi-square test

ADVERSE EVENTS:
Time Frame: Approximately 21 days
Arm/Group | Active Nasal Strip Group | Placebo Nasal Strip Group
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 6/64 | 2/64
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Nasal Strip Group (N=64) | Placebo Nasal Strip Group (N=64)
APPLICATION SITE PRURITUS (General disorders) | 1 (1) | 1 (1)
APPLICATION SITE DISCOLOURATION (General disorders) | 1 (1) | 0 (0)
APPLICATION SITE ERYTHEMA (General disorders) | 0 (0) | 1 (1)
APPLICATION SITE IRRITATION (General disorders) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.